CLINICAL TRIAL: NCT05828004
Title: Effect of Multidisciplinary Team Support on Head and Neck Cancer Patients Receiving Radiotherapy: The SHINE-MDT Randomized Controlled Trial
Brief Title: The SHINE-MDT Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-1831
Record Dates: First submitted 2023-02-02; First posted 2023-04-25 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Carcinoma; Radiotherapy Side Effects
Keywords: Head and Neck Carcinoma; Multidisciplinary Team; Radiotherapy interruption; Supportive Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard care group (No Intervention): The standard care group is the routine care group, that is, under the current standard antitumor treatment and follow-up mode, the patients independently decided whether to carry out nutritional and psychological intervention after the advice from the medical care department of oncology
- MDT care group (Experimental): The MDT care group is the whole-course multidisciplinary care intervention group, which is conducted by a multidisciplinary team composed of the oncology department, nutrition department, mental health center and rehabilitation department.
  Interventions: Behavioral: Whole-Course Multidisciplinary Care Intervention

INTERVENTIONS:
Behavioral: Whole-Course Multidisciplinary Care Intervention — On the basis of standard treatment, all patients were evaluated by senior practice nurses in the Department of Oncology in person at the time of enrollment (before radiotherapy) and once every week during radiotherapy, and once in person/over the phone at 1, 2, 3, and 6 months after radiotherapy.
  Arms: MDT care group

SUMMARY:
Radiotherapy is one of the main treatments for head and neck Carcinoma. The incidence of radiotherapy-related adverse events is greater than 90%, and severe adverse events may lead to the interruption of radiotherapy.

The management of nutritional, psychological, and rehabilitative issues in patients undergoing radiotherapy for head and neck cancer presents unique clinical challenges. We aimed to evaluate the efficacy of the SHINE-MDT (Supportive Holistic Interventions by Nurses and Experts via Multidisciplinary Team) in reducing radiotherapy interruptions and improving patients' quality of life (QoL) compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients had pathologically confirmed malignant head and neck tumors without distant metastasis.
2. Patient age ≥18 years;
3. Patients were scheduled to undergo either postoperative adjuvant radiotherapy or radical radiotherapy, with or without concurrent chemotherapy.
4. Baseline ECOG (Eastern Cooperative Oncology Group) score 0-2;
5. Good cognitive and reading skills, able to complete the questionnaire survey.

Exclusion Criteria:

1. Presence of other malignant tumors aside from head and neck malignancies;
2. A history of prior head and neck radiotherapy;
3. Mental illness or cognitive impairments;
4. Uncontrolled systemic diseases that could significantly affect their QoL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Radiotherapy interruption rate | 5 days
  Interruption of radiotherapy was defined as the actual end date of radiotherapy minus the expected end date at least 5 days

SECONDARY OUTCOMES:
Quality of life score (EORTC QLQ C30) | Weekly during radiotherapy and the first month post-treatment, and at 2, 3, and 6 months post-treatment
  Quality of life score was calculated according to the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 (EORTC QLQ C30)
Quality of life score QLQ-HN35 | Weekly during radiotherapy and the first month post-treatment, and at 2, 3, and 6 months post-treatment
  Quality of life score was calculated according to the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire QLQ-HN35
Nutritional status (NRS 2002, PG-SGA) | Weekly during radiotherapy and the first month post-treatment, and at 2, 3, and 6 months post-treatment
  Nutritional status was calculated according to Nutrition Risk Screening 2002 and Patient-Generated Subjective Global Assessment。
Psychological status (DT, PHQ-9, HADS) | Weekly during radiotherapy and the first month post-treatment, and at 2, 3, and 6 months post-treatment
  Psychological status was calculated according to Distress Thermometer (DT), Hospital Anxiety and Depression Scale (HADS), and Patient Health Questionnaire-9 (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Ph.D, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Pei Y, Wang J, Li J, Chen Y, He J, Wei Z, Liu Z, Su Y, Dai T, Yin L, Deng Y, Zhou J, Tian H, Li Y, Chen X, Zhang S, Chen Y, Yan Q, Li R, Jiang Z, Hu X, Peng X. Multidisciplinary Team Support for Patients With Head and Neck Cancer Receiving Radiotherapy: A Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2547590. doi: 10.1001/jamanetworkopen.2025.47590. PMID 41396606